CLINICAL TRIAL: NCT00936351
Title: Mindfulness as a Rehabilitation Strategy in Schizophrenia
Brief Title: Mindfulness Meditation as a Rehabilitation Strategy for Persons With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4786-W; 0611-01B (Other Grant/Funding Number: VA Rehabilitation Research & Development)
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychotic Disorders
Keywords: schizophrenia; intervention studies; mindfulness meditation; vocational rehabilitation; schizoaffective disorder; psychotic disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Mindfulness; Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Mindfulness Meditation
  Interventions: Behavioral: Mindfulness Meditation
- Arm 2 (Active Comparator): Support Group that involves discussion of work-related issues in which participants are facilitated to assist each other with problem solving and offer support
  Interventions: Behavioral: Support Group (control)

INTERVENTIONS:
Behavioral: Mindfulness Meditation — Mindfulness involves teaching individuals skills that improve their ability to attend to their experience in the present moment while suspending judgment and to purposefully shift their attention. Thus mindfulness enhances the ability to monitor and manage emotions and thought processes so that individuals can reflect on, choose, and implement more effective responses. This intervention has been adapted from mindfulness based stress reduction treatment.
  Arms: Arm 1
Behavioral: Support Group (control) — A support group during which participants can discuss with each other any issues, problems, or successes at work will be conducted as the control portion.
  Arms: Arm 2

SUMMARY:
The purpose of this study is to develop a treatment manual for mindfulness meditation to be taught in a group format to individuals with schizophrenia who are engaged in vocational rehabilitation. This study will also determine whether mindfulness meditation is beneficial in terms of improving work function by reducing distressing emotional states and thinking patterns.

DETAILED DESCRIPTION:
Objectives: Schizophrenia involves numerous difficulties including being aware of ones' own thoughts and tolerating painful affects. As a result, persons with schizophrenia find coping with life stressors quite challenging and thus have difficulty engaging successfully in psychosocial activities such as work in spite of state of the art programs. To address this problem this study will evaluate an intervention that has come to the fore that targets these impairments called mindfulness. Mindfulness involves teaching individuals skills that improve their ability to attend to their experience in the present moment while suspending judgment and to purposefully shift their attention. Thus mindfulness enhances the ability to monitor and manage emotions and thought processes so that individuals can reflect on, choose, and implement more effective responses. Use of mindfulness skills with other populations has led to more sustained behavior change than occurs with standard treatments. Recently research has begun to indicate mindfulness interventions can be delivered with success for individuals with schizophrenia. This pilot study will be a first step in adapting mindfulness as a cognitive intervention for individuals with schizophrenia who are engaging in vocational rehabilitation in order to maintain their functional gains beyond the end of the program. Key questions to be answered through this study include: (1) Can a mindfulness manual be developed that helps persons with schizophrenia enrolled in vocational rehabilitation exhibit better work function and reduced levels of distressing emotional states and thinking patterns?; (2) Can materials necessary for the faithful transmission of the mindfulness group intervention/manual (MGI) in the current study be created?; (3) Can mindfulness skills be adapted and successfully taught to and accepted by persons with schizophrenia in a group setting?: (4) Will individuals with schizophrenia who practice mindfulness benefit?; (5) What are the effect sizes with a reasonable control to study the effectiveness of the manualized MGI? Research Design: This study will take place over 3 years and is divided into two phases: manual development and pilot study. In the manual development phase existing mindfulness protocols will be adapted to target work function of persons with schizophrenia. The randomized controlled pilot study phase will explore the effects of the intervention on key outcome measures.

Methodology: A total of 52 individuals with schizophrenia or schizoaffective disorder will be recruited from the Roudebush VA Medical Center (18 in the non-randomized, non-controlled manual development phase 1 and 34 in the randomized controlled pilot phase 2). In phase one, manual development, 18 participants will be recruited and following informed consent, screened for eligibility using the SCID and anxiety measures. Once enrolled, three successive groups of 6 participants will attend an 8-week mindfulness program consisting of two 60-minute group training and practice sessions each week. The mindfulness program will incorporate didactic and experiential elements aimed at learning mindfulness skills and establishing a daily mindfulness practice. Based on the experience gained working with each of these three initial cohorts, a mindfulness manual will be created. In phase two, the pilot of the mindfulness manual, 34 additional participants will be recruited and randomized to the mindfulness intervention or support group control. All groups will complete assessments at baseline, monthly, at program end and 6 months after program end as well as formative and summative program evaluations.

Clinical Significance: Results of this study will yield materials necessary to begin the process of assembling a body of research validating scientifically the therapeutic value of mindfulness for veterans with schizophrenia who are enrolled in vocational rehabilitation. Findings may ultimately provide the VA system with information regarding a potentially cost effective approach to the care of these veterans who are disabled by a chronic mental illness that would be exportable to other VA vocational rehabilitation programs that have patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* patients with SCID I confirmed DSM-iV diagnosis of schizophrenia or schizoaffective disorder
* in a post acute phase of illness defined by no hospitalizations or changes in type of psychotropic medication or place of residence in the past 30 days
* who are either already enrolled in vocational rehabilitation and working or willing to enroll in vocational rehabilitation and begin working

Exclusion Criteria:

* history of mental retardation
* active substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louanne W Davis, PsyD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Mindfulness Meditation
  Mindfulness involves teaching individuals skills that improve their ability to attend to their experience in the present moment while suspending judgment and to purposefully shift their attention. Thus mindfulness enhances the ability to monitor and manage emotions and thought processes so that individuals can reflect on, choose, and implement more effective responses. This intervention was adapted from Mindfulness-Based Stress Reduction, an 8-week program developed by Jon Kabat-Zinn.
- Arm 2: Support Group
  The support group leader offered empathic statements, support and led discussion of work related issues and concerns, facilitating members to support and help one another with problem-solving.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 18 | 16
Completed | 15 | 14
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Mindfulness Meditation
  Mindfulness involves teaching individuals skills that improve their ability to attend to their experience in the present moment while suspending judgment and to purposefully shift their attention. Thus mindfulness enhances the ability to monitor and manage emotions and thought processes so that individuals can reflect on, choose, and implement more effective responses. This intervention has been adapted from mindfulness based stress reduction treatment.
- Arm 2: Support Group
  Support Group (control): A support group during which participants can discuss with each other any issues, problems, or successes at work will be conducted as the control portion.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Customized [Mean (Standard Deviation); unit: years] | 53.2 (6.1) | 50.1 (10.6) | 51.7 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 17 | 16 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 9 | 21
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Hours
Description: total hours worked over the duration of the 24-week treatment
Time Frame: week 1 through week 24 of treatment
Population: 3 participants were not included due to early dropout
Measure: Mean (Standard Deviation); unit: total hours worked during treatment
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 16 | 15
total hours worked during treatment | 293.5 (40.2) | 234.5 (96.1)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = .04, t-test, 2 sided; Mean Difference (Final Values) = 2.21

2. Primary Outcome: Work Behavior Inventory
Description: The Work Behavior Inventory (WBI: Bryson, et al., 1997) assesses work performance for persons with severe mental illness based on a trained rater's observation of participants at work and an interview with their supervisor. Each of the 35 WBI items are rated as 1- 5 ("persistent problem area" to "frequent area of strength"). The total score is the sum of five sub-scales (social skills, cooperativeness, work habits, work quality, and personal presentation). We divided the total score by 35 to produce a mean score that is conducive to interpretation since there are no established cut-offs for interpretation of the total score. Thus the mean scores range from 1-5 and are interpretable based on the anchors for the likert scale ranging from 1 (persistent problem area" to 5 ("frequent area of strength). Good to excellent interrater reliability was found for raters in this study, with intraclass correlations of .79-.98.
Time Frame: week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 16 | 15
units on a scale | 3.6 (0.4) | 3.0 (0.7)

3. Primary Outcome: Weeks
Description: Vocational rehabilitation staff tracked weekly work hours verified by supervisors and reported the data to study staff during the 24-week interventions. Therefore possible values for total weeks worked range from 1-24.
Time Frame: weeks 1-24
Measure: Mean (Standard Deviation); unit: total number of weeks
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 16 | 15
total number of weeks | 15.2 (1.9) | 12.8 (4.7)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

LIMITATIONS AND CAVEATS:
The sample was middle-aged males with chronic schizophrenia, not representative of the broader population. Raters of work quality were not blinded to condition. Mindfulness and support conditions were not equally matched on intensity of intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No